CLINICAL TRIAL: NCT06945705
Title: A Prospective, Single-arm, Multi-center Clinical Trial of Furmonertinib Combined With Anlotinib as First-line Treatment for Advanced NSCLC With EGFR-sensitive Mutations and Brain Metastasis.
Brief Title: A Clinical Trial of Furmonertinib Combined With Anlotinib as First-line Treatment for Advanced NSCLC With EGFR-sensitive Mutations and Brain Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB-HZ001
Record Dates: First submitted 2025-03-04; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: NSCLC
Keywords: NSCLC; EGFR
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- furmonertinib combined with anlotinib (Experimental): furmonertinib combined with anlotinib
  Interventions: Drug: furmonertinib combined with anlotinib

INTERVENTIONS:
Drug: furmonertinib combined with anlotinib — furmonertinib: 160 mg po qd Anlotinib: 8 mg per day, orally administered.The treatment cycle is every 3 weeks, with each cycle lasting 21 days. Anlotinib are taken on Days 1-14 of each cycle.

SUMMARY:
EGFR mutation-positive NSCLC patients have a higher risk of developing brain metastases. The prognosis is poor for patients presenting with brain or leptomeningeal metastases at any stage, particularly those with such metastases at initial diagnosis, who have the worst prognosis. Furmonertinib, as a novel EGFR-TKI, enhances its lipophilicity by incorporating a trifluoroethoxy pyridine group. Preclinical animal studies further confirm that both Furmonertinib (AST2818) and its metabolite (AST5902) exhibit excellent intracranial distribution. This provides strong theoretical support for the effective treatment of lung cancer brain metastasis patients with Furmonertinib.

EGFR TKI-based combination therapies, as a strategy to delay disease progression, have consistently been a focal point in medical research. Among these, antiangiogenic agents are increasingly recognized for their synergistic effects when combined with TKIs, jointly inhibiting tumor growth, proliferation, and metastasis.Such combinations have demonstrated clear efficacy and manageable safety profiles.

Based on this, the current study aims to explore the efficacy and safety of first-line treatment with 160 mg Furmonertinib combined with anlotinib for advanced NSCLC patients with EGFR-sensitive mutations and brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet all of the following inclusion criteria to be enrolled in this study:

  1. Patients must voluntarily agree to participate in the study and sign a written informed consent form.
  2. Patients must be ≥18 years old, regardless of gender.
  3. Patients must have histologically or cytologically confirmed advanced NSCLC, staged as AJCC TNM 9th edition Stage IV.
  4. Histological or cytological report issued by a hospital or a third-party testing institution recognized by the national assessment confirmed the presence of EGFR 19Del or L858R mutations, with or without other EGFR mutations.
  5. Patients must have an ECOG performance status score of 0-2 and be expected to survive for at least 12 weeks, as determined by the investigator.
  6. Patients must have brain parenchymal metastases confirmed by CT or MRI scans, with or without symptoms (as judged by the investigator).
  7. Patients must have at least one measurable lesion based on RECIST 1.1 criteria.
  8. Patients must not have received prior systemic anticancer therapy for advanced/metastatic NSCLC, including standard chemotherapy, biological therapy, targeted therapy, immunotherapy, or investigational drug therapy. Patients who received adjuvant or neoadjuvant therapy (chemotherapy and/or radiotherapy) are eligible if there has been no disease progression within 6 months of treatment completion. Patients who received local therapy (radiotherapy or pleural perfusion therapy) are also eligible if the treated lesion is not a target lesion.
  9. Patients must meet the following organ function criteria:

     Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L. Platelet count ≥75 × 10⁹/L. Hemoglobin (HGB) ≥80 g/L. Serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN). For patients with liver metastases, TBIL may be up to 3 times ULN. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN.

     For patients with liver metastases, AST and ALT may be up to 5 times ULN. Serum creatinine (SCr) ≤1.5 times ULN, or creatinine clearance rate ≥50 mL/min (calculated using the Cockcroft-Gault formula).
  10. Male patients with reproductive potential and female patients with a possibility of pregnancy must use highly effective contraceptive methods (e.g., oral contraceptives, intrauterine devices, abstinence, or barrier contraception combined with spermicide) during the study and for 12 months after treatment discontinuation.

Exclusion Criteria:

* Patients with any of the following criteria are not eligible for enrollment in this study:

  1. Patients whose diagnosis cannot be confirmed as non-small cell lung cancer (NSCLC) through histological or cytological examination.
  2. Patients who have leptomeningeal metastasis confirmed by MRI and/or positive cerebrospinal fluid (CSF) cytology, but no evidence of brain parenchymal metastasis.
  3. Patients who are expected to require other systemic anticancer therapies outside of this study during the trial period.
  4. Patients with a history of malignancies diagnosed within the past 2 years, excluding well-controlled basal cell carcinoma of the skin, cervical carcinoma in situ, or ductal carcinoma in situ of the breast.
  5. Patients with significant gastrointestinal diseases that may affect drug intake or absorption, including but not limited to peptic ulcers or inflammatory bowel disease.
  6. Patients with known or suspected allergies to the study drugs (furmonertinib and anlotinib) or any components of their formulations.
  7. Patients who have previously received any epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) therapy.
  8. Patients who have used strong CYP3A4 inhibitors or inducers within 7 days before the first dose of the study drug or are expected to require long-term use during the trial. Additionally, patients who have used Chinese herbal medicine or formulations with an antitumor indication within 2 weeks before the first dose or are expected to require such use during the trial.
  9. Patients with a history of interstitial lung disease, drug-induced ILD, or radiation pneumonitis requiring corticosteroid therapy. Patients with acute exacerbation or progressive pulmonary symptoms at baseline, or those deemed unsuitable for enrollment by the investigator due to high-risk factors for ILD, are also excluded.
  10. Patients with significant arrhythmias (e.g., QT interval >470 ms) or heart failure (left ventricular ejection fraction <50%).
  11. Pregnant or breastfeeding women.
  12. Patients who are currently participating in or have participated in other clinical trials within the past 4 weeks.
  13. Patients with severe acute or chronic medical or psychiatric conditions, as judged by the investigator, that may increase the risks associated with participation in the study or interfere with the interpretation of study results. This also includes patients who are unlikely to complete the study or comply with its requirements due to management-related or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2028-10-02 (Estimated)

PRIMARY OUTCOMES:
Safety（Phase One: Safe Introduction Phase） | Up to 6 months
  When subjects receive ≥3 cycles of investigational treatment or discontinue due to intolerable toxicities, safety analysis will commence. If 2 cases of ≥ Grade 3 TRAEs occur, the study will terminate.
progression-free survival (PFS) (Stage Two: Formal Research Phase） | Up to 42 months

SECONDARY OUTCOMES:
objective response rate (ORR)(Stage Two: Formal Research Phase） | Up to 42 months
disease control rate (DCR)(Stage Two: Formal Research Phase） | Up to 42 months
duration of response（DOR）(Stage Two: Formal Research Phase） | Up to 42 months
12m-PFS (Stage Two: Formal Research Phase） | Up to 12 months
18m-PFS(Stage Two: Formal Research Phase） | Up to 18 months
CNS objective response rate（CNS ORR）(Stage Two: Formal Research Phase） | Up to 42 months
CNS disease control rate（CNS DCR）(Stage Two: Formal Research Phase） | Up to 42 months
CNS progression-free survival（CNS PFS）(Stage Two: Formal Research Phase） | Up to 42 months
Safety（Stage Two: Formal Research Phase） | Up to 42 months
  The occurrence rate and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Undecided